CLINICAL TRIAL: NCT05012072
Title: Reductions in Biopsychosocial Risks for Pregnant Latina Women and Their Infants: The Mastery Lifestyle Intervention (MLI)
Brief Title: Reducing Pregnancy Risks: The Mastery Lifestyle Intervention
Acronym: MLI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microgen LLC (Industry)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Roberta Jeanne Ruiz, Research Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2021-07-27; First posted 2021-08-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Wellness 1; Preterm Birth
Keywords: Latina; Pregnancy; Mental Health; Corticotropin Releasing Hormone; Progesterone; Estriol; Gestational age; African American women
MeSH Terms: conditions — Premature Birth; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Usual care group: routine prenatal care by private practice provider Experimental group: Six week group session of the MLI
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The PI will not be allowed to review any data that is not deidentified. The statistician will also not know which participant is in which group by participant names, only by deidentified data.
  The clinical outcomes assessor will not know the group the participant has been in or their study number, but will know the participant names to be able to put the clinical outcomes in the database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLI Experimental group (Experimental): 6 group sessions over 6 weeks with pregnant Latinas and African Americans starting at 14-20 weeks to 21-27 weeks in their prenatal care setting.
  Interventions: Behavioral: The Mastery Lifestyle Intervention
- Control usual prenatal care (No Intervention): Only data collection but no intervention

INTERVENTIONS:
Behavioral: The Mastery Lifestyle Intervention — Combination cognitive behavioral intervention of phase 3 CBT using ACT and PST
  Arms: MLI Experimental group

SUMMARY:
This randomized controlled trial will test an intervention called the Mastery Lifestyle Intervention (the MLI) that was developed from data of 1000+pregnant Hispanic women related to risks of preterm birth. The investigators will deliver a psychoeducational intervention that is manualized over 6 group sessions. The investigators will also have a usual care group that receives standard prenatal care. The investigators plan to enroll 238 pregnant women and start the study with them at 14-20 weeks gestation. The investigators will also test the biological response of the intervention by measuring Corticotropin Releasing Hormone, progesterone, estriol, and test for cotinine. The investigators will also determine any effect on infant outcomes at delivery.

DETAILED DESCRIPTION:
To address the gaps related to interventions for Hispanic Mexican American and African American pregnant women, the investigators have developed and successfully pilot tested the Mastery Lifestyle Intervention (MLI): a culturally-relevant, manualized psychosocial group intervention that integrates two evidence-based behavioral therapies - Acceptance and Commitment Therapy (ACT) and Problem-Solving Therapy (PST). The MLI is a 6-week program designed to be integrated into regular prenatal care to facilitate more comprehensive care delivered by a nurse practitioner (NP) or certified nurse midwife (CNM). We propose the following hypotheses for a randomized controlled trial: Hypothesis 1a: Participants in the 6-week MLI will have decreased depressive symptoms, anxiety, stress, disengaged coping, and increased active coping compared to UC at end-of-treatment and after 6 weeks. Hypothesis 1b: The effects of MLI versus UC on depression, anxiety, stress, acculturative stress, and coping will be mediated via psychological flexibility and moderated by acculturation. Hypothesis 2a: Compared to UC, MLI participants will have significantly lower mean levels of CRH over time from baseline to end-of-treatment. Hypothesis 2b: Compared to UC, MLI participants will have significantly higher progesterone levels and lower estriol levels (higher progesterone/estriol ratios) over time from baseline to end-of-treatment. Hypothesis 3: As compared to UC, infants from mothers in the MLI group will have longer gestational age, greater birth weight, and fewer NICU admissions.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent;
* Ability to read and speak English
* Pregnant at 14-20 weeks gestation with one fetus, intrauterine pregnancy, gestational dating will be reviewed before enrollment via ultrasound administered per standard of care
* Self-identification as African American or Hispanics
* Age 18 to 45 years
* Currently living in the U.S.; Women who identify as just getting along, nearly poor, or poor upon prescreen.
* Women who score 10 or greater on the Center for Epidemiological Studies Depression Scale (CES-D) OR 5 or greater on the Generalized Anxiety Disorder-7 scale (GAD-7), or 14 or > on the Perceived Stress Scale as administered by clinical staff of the participating provider
* Willingness to adhere to the MLI regimen or usual care regimen

Exclusion Criteria:

After initial review of the electronic health record (EHR):

* Major systemic infections such as HIV, hepatitis
* <18 years of age or >45 years of age
* Enrollment in a prenatal program such as the Nurse Family Partnership
* Severe cognitive or psychiatric impairment per judgment of providers, that precludes cooperation with study protocol
* Inability to read English

Women who develop GDM after enrollment in the study will remain in the study. Development of hypertension or preeclampsia, pyelonephritis, or GDM will be considered an effect modifier in analysis of infant outcomes. Current antidepressant use will not be exclusionary and will also be used as an effect modifier. Further rationale for the exclusion criteria is:

* Only singleton pregnancies are included as the mechanisms of PTB are thought to differ with multiples.
* We do not exclude participants based on language (English or Spanish) spoken. We expect heterogeneity in language spoken and expect that there may be women who use both languages. Our prior study findings indicate that the risk of PTB is greatest among English-speaking and bilingual women, although we believe that all women will receive benefit from the MLI.
* Girls <18 are excluded as the intervention is designed to improve emotional wellbeing and quality of life in mature adults; girls <18 may not be cognitively ready for the adult intervention and may need an intervention tailored to their stage of development. Girls under 18 also have a different set of risks than women over 18 years of age.
* We will control the use of progesterone treatment statistically.
* Women who develop gestational diabetes after enrolling in the study will remain in the study.
* At enrollment or during the study, anyone who is prescribed antidepressant or anti-anxiety medications will be eligible for the study. We will make note of it and control it in analysis. If a participant is referred for individual therapy, we will obtain data from the prenatal record and control for that in the analysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Female between 14 to 20 weeks at the time of enrollment.
Enrollment: 238 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Assessing change over time: 14-20 weeks, 21-27 weeks, 32-36 weeks pregnant
  Self Report questionnaire GAD-7
Depression | Assessing change over time:14-20 weeks, 21-27 weeks, 32-36 weeks pregnant
  Self Report questionnaire CES-D
Stress | Assessing change over time:14-20 weeks, 21-27 weeks, 32-36 weeks pregnant
  Self Report questionnaire-PSS
Coping levels | Assessing change over time:14-20 weeks, 21-27 weeks, 32-36 weeks pregnant
  Self Report questionnaire The Brief Cope

SECONDARY OUTCOMES:
To explore the effect of the MLI, versus a usual care group, on the neuroendocrine risk factor of preterm birth (Corticotropin Releasing Hormone (CRH).from baseline to end-of treatment. | Assessing change over time:14-20 weeks gestation, 21-27 weeks gestation
  Corticotropin Releasing Hormone is part of the maternal fetal responses to stress, anxiety, and depressive symptoms.
To explore the effect of the MLI, versus a usual care group, on neuroendocrine risk factors (progesterone) on preterm birth from baseline to end-of treatment. | Assessing change over time:14-20 weeks gestation, 21-27 weeks gestation
  Progesterone is part of the maternal fetal responses to stress, anxiety, and depressive symptoms.
To explore the effect of the MLI, versus a usual care group, on the neuroendocrine risk factor of Estriol. | Assessing change over time:14-20 weeks gestation, 21-27 weeks gestation
  Estriol is part of the maternal fetal response to stress, anxiety, and depressive symptoms.

OTHER OUTCOMES:
To explore the effect of the MLI on infant gestational age at birth | After delivery
  Health outcomes of the infants after usual care or after treatment with the intervention to further determine efficacy.
To explore the effect of the MLI on infant birthweight | After Delivery
  Health outcomes of the infants after usual care or after treatment with the intervention to further determine efficacy.
To explore the effect of the MLI on infants being admitted to the Neonatal Intensive Care Unit | After Delivery
  Health outcomes of the infants after usual care or after treatment with the intervention to further determine efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta J Ruiz, PhD, Principal Investigator — University of Houston
Locations (1):
- Women's Specialist of PLLC, Webster, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz RJ, Grimes K, Spurlock E, Stotts A, Northrup TF, Villarreal Y, Suchting R, Cernuch M, Rivera L, Stowe RP, Pickler RH. The mastery lifestyle intervention to reduce biopsychosocial risks for pregnant Latinas and African Americans and their infants: protocol for a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Dec 28;22(1):979. doi: 10.1186/s12884-022-05284-9. PMID 36577949
- [Result] Ruiz RJ, Newman M, Records K, Wommack JC, Stowe RP, Pasillas RM. Pilot Study of the Mastery Lifestyle Intervention. Nurs Res. 2019 Nov/Dec;68(6):494-500. doi: 10.1097/NNR.0000000000000384. PMID 31693556
- See also: PubMed — http://pubmed.ncbi.nlm.nih.gov/31693556/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT05012072/Prot_SAP_ICF_002.pdf